CLINICAL TRIAL: NCT02295618
Title: Can the ETView VivaSight SL Rival the Macintosh Laryngoscopy With Conventional Tube During Adult Resuscitation by Novice Physicians: a Randomized Crossover Simulation Study.
Brief Title: ETI During Intubation
Acronym: SL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ETI/2014/41
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Intubation; Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ETI with chest compressions (Experimental): endotracheal intubation (ETI) during child mannikin resuscitation with uninterrupted chest compressions. In order to simulate the difficulties associated with intubation during uninterrupted chest compressions, CPR was performed by using LUCAS-2 (Physio-Control, Redmond, WA, U.S.).
  Interventions: Device: Standard tracheal tube; Device: ETView VivaSight SL
- ETI without chest compressions (Experimental): Endotracheal intubation of child mannikin during resuscitation without chest compressions.
  Interventions: Device: Standard tracheal tube; Device: ETView VivaSight SL

INTERVENTIONS:
Device: Standard tracheal tube — Intubation using Macintosh laryngoscope and standard tracheal tube
Device: ETView VivaSight SL — Intubation using ETView VivaSight SL

SUMMARY:
The objective of this study is to compared effectiveness of intubation using ETView VivaSight SL and standard tracheal tube during resuscitation performed by a novice-physicians.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* maximum 1 year of work experience in medicine
* maximum 10 clinical intubations

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2014-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Time to intubation | 1 day
  time from insertion of the blade to the first manual ventilation of the manikin´s lungs. If time of intubation is over than 60 seconds, attempt was recognized as failure.

SECONDARY OUTCOMES:
Success of intubation | 1 day
  effectiveness of the first, second and third intubation attempts and overall effectiveness of intubation by participants using four intubation devices. If the examinee failed at all attempts, the case was excluded from the time calculations.
Cormack-Lehan scale | 1 day
  self reported Cormack-Lehan scale during intubation

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — Institute of Cardiology
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland

REFERENCES:
- [Derived] Kurowski A, Szarpak L, Truszewski Z, Czyzewski L. Can the ETView VivaSight SL Rival Conventional Intubation Using the Macintosh Laryngoscope During Adult Resuscitation by Novice Physicians?: A Randomized Crossover Manikin Study. Medicine (Baltimore). 2015 May;94(21):e850. doi: 10.1097/MD.0000000000000850. PMID 26020389